CLINICAL TRIAL: NCT07093437
Title: Dispositivos Adhesivos Frente a Dispositivos elásticos Para la sujeción de la Sonda Urinaria en el Paciente crítico Estudio Experimental
Brief Title: Adhesive Devices Versus Elastic Devices for Urinary Catheter Securement in Critically Ill Patients Experimental Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Hospital de la Santa creu i Sant Pau - Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIBSP-DAE-2025-22; SLT035/24/000015 (Other: Generalitat de Catalunya)
Record Dates: First submitted 2025-07-09; First posted 2025-07-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Pressure Injuries; Pain; Catheter-Associated Urinary Tract Infection; Medical Device Site Injury
Keywords: Urinary catheter securement; Urinary catheter fixation; Catheter-associated urinary tract infections; pain; Meatal pressure injuries
MeSH Terms: conditions — Pressure Ulcer; Pain | interventions — Urinary Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urinary catheter securement with adhesive device (Experimental): * Site of catheter securement: The urinary catheter will be secured on the anterior aspect of the thigh. The exact placement site will be chosen with the patient's leg bent, to ensure that the securement allows for future leg movement without causing tension or pulling on the catheter.
  * Catheter anchoring method: In female patients, the catheter will be anchored at the "Y" junction of the urinary catheter. In male patients, since the external portion of the catheter is shorter, the anchoring will be done just after the sampling port of the urine collection system.
  * Skin protection: Before applying the adhesive, a protective barrier spray (Cavilon® spray, 3M) will be applied to the selected skin area to prevent potential skin injury
  * Application: The device will be applied following the manufacturer's instructions.
  * Replacement: The device will be changed every 72 hours or sooner if needed. The thigh used for securement will be alterned at every change.
  Interventions: Device: GRIP-LOK FOLEY SECUREMENT DEVICE ®
- Urinary catheter securement with elastic device (Experimental): * Site of catheter securement: The urinary catheter will be secured on the anterior aspect of the thigh. The exact placement site will be selected with the patient's leg bent, to ensure that the securement allows for subsequent leg movement without causing pulling or tension on the catheter.
  * Catheter anchoring method: In female patients, the catheter will be anchored at the "Y" junction of the urinary catheter. In male patients, since the external portion of the catheter is shorter, the anchoring will be done just after the sampling port of the urine collection system.
  * Skin protection: The elastic band will be adjusted appropriately to minimize catheter movement while allowing normal blood circulation in the limb.
  * Application: The device will be applied following the manufacturer's instructions.
  * Replacement:The device will be changed every 72 hours, or sooner if necessary. The thigh used for securement will be alternated at every change
  Interventions: Device: CONVEEN, ELASTIC LEG WRISTBAND FOR URINARY CATHETER

INTERVENTIONS:
Device: GRIP-LOK FOLEY SECUREMENT DEVICE ® — * Used device: adhesive
  * Specific Skin protection: with non alcohol barrier film
  Arms: Urinary catheter securement with adhesive device
Device: CONVEEN, ELASTIC LEG WRISTBAND FOR URINARY CATHETER — The elastic wristband will be adjusted appropriately to minimize catheter movement while allowing normal blood circulation in the limb.
  Arms: Urinary catheter securement with elastic device

SUMMARY:
Nowadays there are two types of urinary catheter securement devices, adhesive and elastic bands. The goal of this clinical trial is to determine which type of device-adhesive or elastic-is more effective for securing urinary catheters in critically ill patients. The study also aims to evaluate the prevention of urethral meatus injuries, patient discomfort, and the incidence of catheter-associated urinary tract infections .

The main questions the trial aims to answer are:

* Which device type better prevents injuries to the urethral meatus?
* Which device reduces discomfort for patients?
* Which device lowers the incidence of catheter-associated urinary tract infections?

Participants will:

* Use either an adhesive or an elastic device to secure their urinary catheter during their stay in critical care
* Be monitored regularly to assess any injuries, discomfort, or infections related to the catheter
* Provide feedback on their comfort and any complications experienced, if they are able to communicate

DETAILED DESCRIPTION:
Urinary catheters (UC) are commonly used medical devices in Intensive Care Units (ICU), Between 50 % and 80 % of ICU patients have a UC in place. Although this is a relatively simple device, it is not free from risks, and complications associated with its use can be diverse and potentially serious.

Among the most relevant complications are three. First, catheter-associated urethral meatus injuries, which are lesions caused by continuous pressure from the catheter on surrounding tissues, affecting the glans, penis, or labia minora. The prevalence of these injuries in critically ill patients ranges between 13 % and 36 %. Secondly, pain and discomfort, occurring in approximately 47 % of UC users. Thirdly, catheter-associated urinary tract infection (CAUTI) is a frequent complication; in Spanish ICUs, it has accounted for 25 % to 30 % of all device-associated infections in recent years.

Securing urinay catheter to the leg is recommended by several international clinical practice guidelines (CPG) to prevent complications associated with UC use. In Spain, the national ITU ZERO initiative-led by the Ministry of Health and the Spanish Society of Intensive and Coronary Care Nursing-includes catheter securement as part of recommended care to reduce the risk of UC-related UTIs in critically ill patients.

Recent studies have evaluated the effectiveness of thigh securement of UC in ICU patients. One 2024 study showed that secured catheters significantly reduced the incidence of meatal injuries, decreased associated discomfort and lowered the risk of CAUTI.

Nowadays, two main types of commercial catheter securement devices are available: elastic wristband-style devices and adhesive-based devices. However, recent studies have not directly compared the effectiveness of these two types, and expert opinions vary.

Moreover, CPG recommend securement devices but do not specify which method is best for critically ill patients. This lack of clear guidelines and robust scientific evidence has resulted in low adherence to catheter securement practices among nurses. Prevalence studies from Canada and the UK (2016) reported low adherence rates. A recent qualitative study concluded that this low adherence stemmed from lack of training, ambiguous recommendations, limited scientific evidence, and insufficient engagement of nursing staff in care research.

In conclusion, urinary catheter securement in critically ill patients is a fundamental intervention for preventing complications, yet there remains a clear lack of comparative evidence between available devices, limiting professionals' ability to select the safest and most effective option. This knowledge gap justifies the need for research to determine which of the two securement types-adhesive or elastic-is more beneficial in this patient population.

________________________________________ Hypothesis: In critically ill patients, urinary catheter securement using adhesive devices is more effective than elastic wristband-style devices in preventing urethral meatus injuries, reducing discomfort, and decreasing the incidence of catheter-associated urinary tract infections.

It is proposed that adhesive devices provide greater stability and exert less pressure on tissues, thereby reducing iatrogenic complication risk and improving patient well-being, compared with elastic devices that may cause vascular compromise or skin irritation in edematous or fragile-skin patients.

This hypothesis will be tested by comparing both securement methods in terms of incidence of injuries, pain, and urinary tract infections in critically ill patients requiring long-term urinary catheters.

________________________________________ OBJECTIVES

Primary Objective:

To evaluate and compare the effectiveness of adhesive versus elastic wristband securement devices for urinary catheters in preventing catheter-associated complications in critically ill patients.

Secondary Objectives:

* Compare the effectiveness of adhesive versus elastic securement in preventing urethral meatus injuries in critically ill patients.
* Evaluate the effect of adhesive versus elastic securement on reducing discomfort and pain related to catheter use in critically ill patients able to communicate.
* Compare the incidence of catheter-associated urinary tract infections between groups using adhesive versus elastic securement devices.
* Analyze patient perceptions and experiences (in communicative patients) regarding the two types of securement devices.
* Identify and describe adverse events related to securement device use, such as catheter obstruction, skin lesions, and accidental catheter dislodgment.

METHODOLOGY This study will be conducted in the Intensive Care Unit (ICU) of Hospital de la Santa Creu i Sant Pau. It is an experimental, randomized, open-label trial with two intervention groups. Group 1 (G1) patients will receive urinary catheter securement using a commercially available adhesive device, while Group 2 (G2) patients will use an elastic wristband device. In this study, patients will be randomly assigned to G1 or to G2.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Pacients with an urinary catheter inserted within the past 24 hours
* Expected duration of catheterization >48 hours
* Estimated ICU lenght os stay > 48 hours

Exclusion Criteria:

* Known allergy to adhesive tape
* Patients with lesions at the urinary meatus, ongoing urinary tract infection or suspected infection
* Presence of urological or prostatic pathology
* Any condition that prevents securing the urinary catheter to the thigh, such as wounds, burns, or amputations

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Urinary Catheter-related Meatal pressure injuries incidence | Through study completion, an average of 10 days
  Urinary Catheter-related Meatal pressure injuries are localized damage to the skin and underlying tissues around the urinary meatus resulting from continuous mechanical pressure from the catheter. This pressure can impair blood flow, leading to tissue ischemia, breakdown, and ulceration at the site where the catheter contacts the meatus.
Urinary catheter-related pain in comunicative patients incidence | Through study completion, an average of 10 days
  Urinary catheter-related pain refers to the discomfort or pain experienced by patients as a direct consequence of the presence and use of an indwelling urinary catheter. This pain can arise from mechanical irritation of the urethral mucosa, bladder spasms, inflammation of the urinary tract, and tissue trauma during catheter insertion or prolonged use.
  This outcome will be measured only in patients with the ability to communicate effectively. To asses pain severity the Numeric Rating Scale (NRS) will be used. It consists of a scale from 0 to 10, where 0 means no pain and 10 means the worst possible pain. Patients will be asked to rate their current pain by choosing a number that best represents their pain level.
Catheter associated-urinary tract infection incidence | Through study completion, an average of 10 days
  Catheter-Associated Urinary Tract Infection (CAUTI) is a type of urinary tract infection that occurs in patients who have an indwelling urinary catheter. It is caused by the introduction and colonization of microorganisms, often bacteria, along the catheter into the urinary tract.

CONTACTS AND LOCATIONS:
Overall Officials: Neus Calpe Damians, PhD, Study Director — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Institut de Recerca Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Data sharing is not planned due to limitations in consent obtained from participants. Moreover, the dataset is proprietary and sharing is restricted by institutional policies.

REFERENCES:
- [Background] Shenhar C, Mansvetov M, Baniel J, Golan S, Aharony S. Catheter-associated meatal pressure injury in hospitalized males. Neurourol Urodyn. 2020 Jun;39(5):1456-1463. doi: 10.1002/nau.24372. Epub 2020 Apr 27. PMID 32339318
- [Background] Jang EB, Hong SH, Kim KS, Park SY, Kim YT, Yoon YE, Moon HS. Catheter-Related Bladder Discomfort: How Can We Manage It? Int Neurourol J. 2020 Dec;24(4):324-331. doi: 10.5213/inj.2040108.054. Epub 2020 Dec 31. PMID 33401353
- [Background] Wound Ostomy and Continence Care Nurses society. Indwelling Urinary Catheter Securement: Best Practice for Clinicians. WOCNS, USA;2012.
- [Background] Calpe-Damians N, Wennberg-Capellades L, Ventura-Rosado A, Gonzalez-Engroba R, Enriquez-Perez N, Vicario-Martos C, Roldos-Gales A, Guri-Lopez T, Rafart-Aguado S, Ramirez-Ramon A, Llaurado-Serra M. Effectiveness and safety of a simple catheter securement device aimed at preventing catheter-associated urinary tract infection in intensive care unit patients: A randomized controlled trial. Nurs Crit Care. 2024 Nov;29(6):1788-1798. doi: 10.1111/nicc.13111. Epub 2024 Jul 2. PMID 38955490
- [Background] Holroyd S. The importance of indwelling urinary catheter securement. Br J Nurs. 2019 Aug 8;28(15):976-977. doi: 10.12968/bjon.2019.28.15.976. No abstract available. PMID 31393768
- [Background] Calpe-Damians N, Llaurado-Serra M, Wennberg-Capellades L. Knowledge and beliefs of intensive care nurses about urinary catheter securement: Results of a national survey. Intensive Crit Care Nurs. 2024 Apr;81:103572. doi: 10.1016/j.iccn.2023.103572. Epub 2023 Nov 16. PMID 37977003

DOCUMENTS (2):
  • Statistical Analysis Plan (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT07093437/SAP_000.pdf
  • Informed Consent Form (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT07093437/ICF_001.pdf